CLINICAL TRIAL: NCT05197517
Title: A Randomized, Single-Dose, Two-Way Crossover, Open-Label, Bioequivalence Study of the Two Different Products Containing 10 mg Film Coated Tablet After Oral Administration to 38 Healthy Adult Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Rosuvastatin in Healthy Volunteers Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rania Mahmoud Mohamed (Other)
Collaborators: Future University in Egypt (Other)
Responsible Party: Sponsor-Investigator, Rania Mahmoud Mohamed, Unit director at FRC, Future University in Egypt
Organization: Future University in Egypt (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: VIN-B-20-026
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Bioequivalence
Keywords: Rosuvastatin; Bioequivalence; Randomized; Cross-Over
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: A Randomized, Single-Dose, Two-Way Crossover, Open-Label, Bioequivalence Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin 10 mg film coated tablets (Experimental): Single oral dose of 1 tablet (10 mg)
  Interventions: Drug: Rosuvastatin 10 mg
- Crestor® 10 mg film coated tablets (Active Comparator): Single oral dose of 1 tablet (10 mg)
  Interventions: Drug: Rosuvastatin 10 mg

INTERVENTIONS:
Drug: Rosuvastatin 10 mg — Film Coated Tablets products containing 10 mg Rosuvastatin

SUMMARY:
The present study is conducted to evaluate and compare the relative bioavailability for Rosuvastatin in two different products containing 10 mg film coated tablet after single oral administration.

DETAILED DESCRIPTION:
A Randomized, Single-Dose, Two-Way Crossover, Open-Label, Bioequivalence Study of the two different products containing 10 mg film coated tablet after oral administration to 38 healthy adult volunteers under fasting conditions. Blood samples were collected at different time intervals and stored at -70⁰C freezer. Plasma concentrations of Rosuvastatin were analyzed and determined using a validated LC-MS-MS method then pharmacokinetics and statistical analysis were performed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained for study.
* Age 18 - 55 years,
* Body mass index between 18.5 and 30 kg/m2
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination.
* Vital signs without significant deviations.
* All laboratory screening results are within the normal range or clinically non-significant

Exclusion Criteria:

* History or presence of any disorder or condition that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the investigator.
* History of any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, allergic, dermatologic, hematologic, neurologic, or psychiatric disease, or cancer.
* Any confirmed significant allergic reactions against any drug, or multiple allergies.
* Clinically significant illness 28 days before study phase I.
* Alcohol or any solvent intake.
* Regular use of medication.
* Positive urine screening of drugs of abuse.
* Use of any systemic medications (prescription medications, OTC products, supplements, or herbal preparations) for 14 days prior to dosing and during the study.
* History or presence of significant smoking (more than one pack per day cigarettes) or refusal to abstain from smoking for 48 hours before dosing until checkout.
* Blood donation within the past 60 days.
* Participation in another bioequivalence study within 60 days prior to the start of phase I of the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Pre-dose and 0.5, 1, 2, 2.5, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 6, 7, 10, 12, 24, 48, and 72 hours
  Cmax is observed as the maximum of Rosuvastatin peak concentration
Area under the plasma concentration curve from administration to last observed concentration at time t (AUC(0-t)) | Pre-dose and 0.5, 1, 2, 2.5, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 6, 7, 10, 12, 24, 48, and 72 hours
  The AUC (0-t) is the area under the plasma concentration versus time curve from time zero (predose) to time of last quantifiable concentration (tlast).
Area under the plasma concentration curve extrapolated to infinite time (AUC(0-inf)) | Pre-dose to infinite time
  AUC(0-inf) "the area under the curve," which is a way of measuring the total amount of the active drug in a subject's system over a period of time from administration ("0") to the time that the drug is no longer present in the subject's body ("infinity")

SECONDARY OUTCOMES:
Maximum time (Tmax) | Pre-dose and 0.5, 1, 2, 2.5, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 6, 7, 10, 12, 24, 48, and 72 hours
  Time until Cmax is reached
Elimination Rate Constant (Kel) | Pre-dose and 0.5, 1, 2, 2.5, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 6, 7, 10, 12, 24, 48, and 72 hours
  Kel is a value used in pharmacokinetics to describe the rate at which a drug is removed from the human system
Plasma concentration half-life (t1/2) | Pre-dose and 0.5, 1, 2, 2.5, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 6, 7, 10, 12, 24, 48, and 72 hours
  t1/2 is the time taken for the plasma concentration of a drug to reduce to half its original value. It is used to estimate how long it takes for a drug to be removed from your body.

CONTACTS AND LOCATIONS:
Locations (1):
- Future Research Center (FRC), Cairo, Egypt